CLINICAL TRIAL: NCT01333969
Title: The Effect of Ischemic Preconditioning on Postoperative Pain After Total Knee Arthroplasty, a Randomized, Controlled Trial
Brief Title: Ischemic Preconditioning in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2012-038
Record Dates: First submitted 2011-04-11; First posted 2011-04-12 (Estimated); Results first posted 2024-09-23 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-05

CONDITIONS: Total Knee Arthroplasty; Ischemic Preconditioning; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ischemic Preconditioning

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ishcemic Preconditioning (Active Comparator): In the study group, the patients' operative limb will be preconditioned by inflating the tourniquet for 5 minutes, followed by deflation and a 5-minute reperfusion period. Subsequently, the tourniquet will be inflated for the entire length of the operation (before skin incision to after insertion of the final components).
  Interventions: Procedure: Ischemic Preconditioning
- Control (No Intervention): In the control group, the tourniquet will be used for the entire length of the operation without a preconditioning phase.

INTERVENTIONS:
Procedure: Ischemic Preconditioning — In the study group, the patients' operative limb will be preconditioned by inflating the tourniquet for 5 minutes, followed by deflation and a 5-minute reperfusion period. Subsequently, the tourniquet will be inflated for the entire length of the operation (before skin incision to after insertion of the final components). In the control group, the tourniquet will be used for the entire length of the operation without a preconditioning phase.
  Arms: Ishcemic Preconditioning

SUMMARY:
The application of a tourniquet for 5 minutes and subsequent reperfusion before actual inflation of the tourniquet for total knee arthroplasty (ischemic preconditioning) decreases the level of local inflammation and therefore postoperative pain in response to reperfusion of the ischemic extremity.

DETAILED DESCRIPTION:
During knee surgery your surgeon routinely uses a device called a tourniquet that allows us to temporarily cut of blood supply to the site of surgery. This helps to reduce blood loss and improves operating conditions. When allowing blood back into your leg at the end of the procedure, debris (bone, fat, tissue breakdown products and cement from the surgery) gets washed out and gains access to the rest of your body. In the vast majority of cases this event bares no major clinical consequences, but can rarely result in signs of inflammation of various body systems. Patients with evidence of impaired organ system function such as pre-existing lung and heart disease may be more vulnerable. Previous studies suggest that cutting off the blood supply for a short period of time just before a prolonged episode, could lead to a decrease in the extent of tissue breakdown products in this extremity and may thus be associated with a decrease in the inflammation of other organ systems. We propose to study this theory in knee surgery patients by looking at levels of markers of inflammation present in the blood before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing primary total knee arthroplasty

Exclusion Criteria:

* Patients who chronically use narcotics (<1 month).
* Patients with contraindications (severe peripheral vascular disease, presence of femoral-popliteal bypass grafts, etc.) or no plan for tourniquet use as determined by the clinical care team.
* Patients who are on corticosteroids prior to their surgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stavros G. Memtsoudis, MD, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Result] Memtsoudis SG, Stundner O, Yoo D, Gonzalez Della Valle A, Boettner F, Bombardieri AM, Jules-Elysee K, Poultsides L, Ma Y, Sculco TP. Does limb preconditioning reduce pain after total knee arthroplasty? A randomized, double-blind study. Clin Orthop Relat Res. 2014 May;472(5):1467-74. doi: 10.1007/s11999-013-3106-4. PMID 23761178

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ishcemic Preconditioning | Control
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ishcemic Preconditioning | Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Age | 66.5 [55.7 to 77.3] | 72.5 [59.2 to 85.8] | 70.8 [55.7 to 85.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 33
  Male | 11 | 16 | 27

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain at Rest and Exercise as Assessed by Visual Analogue Scale (VAS) Scores at 48h After Surgery
Description: Visual Analogue Scale (VAS) are used to measure the intensity of pain. The total scale ranged from 0 (no pain) to 10 (excruciating pain). The average value at POD 48hours was reported for each arm/group.
Time Frame: 48hrs after surgery
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ishcemic Preconditioning | Control
Number analyzed (Participants) | 30 | 30
score on a scale
  VAS score at rest | 1.75 [.02 to 2.25] | .71 [.02 to 1.40]
  VAS score with exercise | 3 [1.80 to 4.2] | 1.38 [.44 to 2.32]
Statistical Analysis 1: Comparison: Ishcemic Preconditioning vs Control; Test type: Superiority; p = .043, GEE; Regression analysis using the generalized estimating equations (GEE) method to compare the changes over time in VAS scores at rest and with exercise; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.40 to -0.02]

2. Secondary Outcome: Overall Epidural Volume
Description: Postoperative pain management included an epidural infusion of 10mcg/ml bupivacaine 0.06%/hydromorphone with a basal rate of 4 mL, a demand dose of 4 mL, and a lockout of 10 minutes. Basal rates were reduced to 2 mL and 0 mL in the morning of postoperative Days 1 and 2, respectively and epidural catheters removed on postoperative Day 2. Overall epidural volume was the total volume given over 48 hours.
Time Frame: At 48hrs after surgery
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Ishcemic Preconditioning | Control
Number analyzed (Participants) | 30 | 30
mL | 140.5 (68.4) | 160.8 (70.1)
Statistical Analysis 1: Comparison: Ishcemic Preconditioning vs Control; Test type: Other; p = .043, t-test, 2 sided; Mean Difference (Final Values) = .043

3. Secondary Outcome: Muscle Oxygenation Over Calf at 48h After Surgery
Description: muscle tissue oxygenation was measured using a novel noninvasive near infrared spectroscopy device at baseline and at 48 hours postoperatively
Time Frame: At 48 hrs after surgery
Measure: Mean (Standard Deviation); unit: percentage of muscle tissue
Arm/Group | Ishcemic Preconditioning | Control
Number analyzed (Participants) | 30 | 30
percentage of muscle tissue | 75 (22.4) | 69 (18.5)
Statistical Analysis 1: Comparison: Ishcemic Preconditioning vs Control; Test type: Superiority; p = .584, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = .584

4. Secondary Outcome: Levels of Interleukin 6 (IL6) in Drainage Fluid at 24hr Postoperatively
Time Frame: At 24 hours postoperatively
Population: IL-6 levels could not be measured for all patients.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Groups:
- Ischemic Preconditioning - IL6 Levels: In the study group, the patients' operative limb will be preconditioned by inflating the tourniquet for 5 minutes, followed by deflation and a 5-minute reperfusion period. Subsequently, the tourniquet will be inflated for the entire length of the operation (before skin incision to after insertion of the final components).
- Control - IL6 Levels: In the control group, the tourniquet will be used for the entire length of the operation without a preconditioning phase.
Arm/Group | Ischemic Preconditioning - IL6 Levels | Control - IL6 Levels
Number analyzed (Participants) | 24 | 28
pg/ml | 3.79 [2.4 to 6.6] | 3.57 [2.3 to 7.4]
Statistical Analysis 1: Comparison: Ischemic Preconditioning - IL6 Levels vs Control - IL6 Levels; Test type: Superiority; p = 0.763, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.763

5. Secondary Outcome: Periarticular Circumference of the Knee at 6h, 24h, and 48h
Description: Periarticular circumference of the knee as compared to contralateral side as crude marker of swelling at 6h, 24, and 48h postoperatively. The data from the specified time points (6h, 24h, and 48h) were combined and the average value was reported for each arm/group.
Time Frame: measured at 6 hours, 24 hours, and 48 hours
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Ishcemic Preconditioning | Control
Number analyzed (Participants) | 30 | 30
cm | 2.3 (3.2) | 1.5 (1.1)
Statistical Analysis 1: Comparison: Ishcemic Preconditioning vs Control; Test type: Superiority; p = .602, GEE; Regression analyses based on the generalized estimating equations (GEE) method; Mean Difference (Final Values) = .602

6. Secondary Outcome: Hospital Length of Stay
Time Frame: Up to discharge date
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Ishcemic Preconditioning | Control
Number analyzed (Participants) | 30 | 30
hours | 100.6 [56.2 to 145] | 99.4 [63.4 to 135.4]
Statistical Analysis 1: Comparison: Ishcemic Preconditioning vs Control; Test type: Superiority; p = .8656, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = .8656

7. Secondary Outcome: Physical Therapy Milestone
Description: Amount of time until patients reached their physical therapy milestone (40 ft ambulation) during admission
Time Frame: Up to discharge date
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Ishcemic Preconditioning | Control
Number analyzed (Participants) | 30 | 30
days | 2.0 [1.0 to 3.0] | 3.0 [2.0 to 4.0]
Statistical Analysis 1: Comparison: Ishcemic Preconditioning vs Control; Test type: Superiority; p = .8422, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = .8422

8. Secondary Outcome: Levels of Leukocytes in Drainage Fluid at 24hr Postoperatively
Time Frame: 24 hours postoperatively
Population: some patients were lost to follow up.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Groups:
- Ischemic Preconditioning - Leukocytes: In the study group, the patients' operative limb will be preconditioned by inflating the tourniquet for 5 minutes, followed by deflation and a 5-minute reperfusion period. Subsequently, the tourniquet will be inflated for the entire length of the operation (before skin incision to after insertion of the final components).
- Control - Leukocytes: In the control group, the tourniquet will be used for the entire length of the operation without a preconditioning phase.
Arm/Group | Ischemic Preconditioning - Leukocytes | Control - Leukocytes
Number analyzed (Participants) | 23 | 25
cells/mm^3 | 2487 (2415.74) | 2038 (1778.74)
Statistical Analysis 1: Comparison: Ischemic Preconditioning - Leukocytes vs Control - Leukocytes; Test type: Superiority; p = .526, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = .526

9. Secondary Outcome: Levels of TNF-alpha in Drainage Fluid at 24hr Postoperatively
Time Frame: 24 hours postoperatively
Population: some patients were lost to follow up.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Groups:
- Ischemic Preconditioning - TNF-alpha: In the study group, the patients' operative limb will be preconditioned by inflating the tourniquet for 5 minutes, followed by deflation and a 5-minute reperfusion period. Subsequently, the tourniquet will be inflated for the entire length of the operation (before skin incision to after insertion of the final components).
- Control - TNF-alpha: In the control group, the tourniquet will be used for the entire length of the operation without a preconditioning phase.
Arm/Group | Ischemic Preconditioning - TNF-alpha | Control - TNF-alpha
Number analyzed (Participants) | 28 | 29
pg/ml | 3.72 [3.09 to 4.65] | 3.76 [3.05 to 5.82]
Statistical Analysis 1: Comparison: Ischemic Preconditioning - TNF-alpha vs Control - TNF-alpha; Test type: Superiority; p = .526, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = .526

ADVERSE EVENTS:
Arm/Group | Ishcemic Preconditioning | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes